CLINICAL TRIAL: NCT04094441
Title: Implementation of Data From Pulmonary Function Tests Supervising a Session of Respiratory Physiotherapy of Cystic Fibrosis Children in the VirtualChest Model
Brief Title: Modeling of Chest Physiotherapy Using Impedance Measurements (PHYSIOMOD)
Acronym: PHYSIOMOD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: N° IDRCB: 2017-A02426-47
Record Dates: First submitted 2019-08-19; First posted 2019-09-19 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2019-08

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: one arm, the interventional design is related to additional pulmonary function tests
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- additional pulmonary function tests (Experimental): additional pulmonary function tests
  Interventions: Other: chest physiotherapy

INTERVENTIONS:
Other: chest physiotherapy — chest physiotherapy

SUMMARY:
"The usefulness of respiratory physiotherapy and its execution modalities remains highly debated even though reviews of the literature show that respiratory physiotherapy is able to improve the drainage of bronchial secretions and pulmonary function tests during cystic fibrosis in periods of stability. Different physiotherapy techniques have been developed but the choice of one or the other facing a patient can not currently be recommended. The VirtualChest project, supported by a grant from the National Agency for Research (ANR), aims to develop and validate a physical model of respiratory physiotherapy (6 stages including model establishment pulmonary: bronchial tree and pulmonary mechanics and parietal [steps 1 and 3], a model of mucus [step 2] and modeling the effect of physiotherapy [step 5]). This project is integrated with stages 3 and 5 of this broad project and aims to get on a limited number of children with cystic fibrosis a proof of concept (prediction of drainage efficiency) and especially to feed the proposed physical models in order to subsequent optimization of the model (step 6). The choice cystic fibrosis of the child was justified by the effect demonstrated respiratory physiotherapy, particularly on respiratory functional criteria, and the fact that the parietal mechanics varies physiologically at this age."

DETAILED DESCRIPTION:
"The clinical study will consist in carrying out, before and after hospital respiratory physiotherapy, a measure impedance of the respiratory system by forced oscillations (IOS, impulsometry: measurement during tidal breathing) and a measurement anatomical dead space (duration of the two measurements: 10 minutes). The physiotherapist will make an initial diagnosis (degree of bronchial obstruction), fill a form describing the modalities of the physiotherapy session (methods used) and will evaluate the sputum volume got. On a limited number of children (n = 6), expiratory flow will be measured during the session of physiotherapy ; these measures will be carried out in hypersecreting children able to support a face mask during the session and having had or before have a chest CT scan within 6 months. The objective is to establish a correlation between sputum volume and the degree of improvement of functional respiratory parameters, to establish criteria of central and / or peripheral effect of physiotherapy (""simple"" modeling obtained from measurements impedance of the respiratory system) and to obtain the flow rates necessary and sufficient to mobilize bronchial secretions. The data from this phase will allow to fuel the ""complex"" physical model (distribution mucus in the airways). Moreover, for each of the patients will be recovered the possible scanner performed within ± 6 months of the physiotherapy session which will allow the extraction of the morphology of the airways of the patient. The goal is to get in at least 6 patients a specific morphology of the airways and determine if this morphology implementation allows to improve the model compared to the use of generic modeling or airway tree. A total of 30 elderly Cystic Fibrosis children at least 4 years will be prospectively included."

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of cystic fibrosis
* Physiotherapy session is programmed

Exclusion Criteria:

-

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2019-01-10 (Actual); Primary Completion 2021-01-10 (Actual); Study Completion 2021-01-10 (Actual)

PRIMARY OUTCOMES:
Impedance measurements will be obtained before and after chest physiotherapy using the Impulse Oscillometry System. | 2 hours
  Impedance of the respiratory system: Z5Hz, Z10Hz, Z20Hz, Z35Hz, R5Hz (respiratory system resistance), X5Hz (respiratory system reactance), R5-20Hz (difference R5 - R20Hz)

CONTACTS AND LOCATIONS:
Overall Officials: Christophe Delclaux, PhD, Principal Investigator — APHP
Locations (1):
- Robert Debre Hospital, Paris, France

REFERENCES:
- [Background] Bokov P, Gerardin M, Brialix G, Da Costa Noble E, Juif R, Foucher AV, Le Clainche L, Houdouin V, Mauroy B, Delclaux C. Beneficial short-term effect of autogenic drainage on peripheral resistance in childhood cystic fibrosis disease. BMC Pulm Med. 2022 Jun 21;22(1):241. doi: 10.1186/s12890-022-02039-2. PMID 35729620